CLINICAL TRIAL: NCT05432024
Title: Evaluation of Ablation Lesions Using Cardiovascular Magnetic Resonance Imaging
Acronym: ENABLE-CMR
Status: Recruiting | Type: Observational
Sponsor: R&D Cardiologie (Other)
Responsible Party: Principal Investigator, L.V.A. Boersma, Clinical professor, R&D Cardiologie
Other Study IDs: RDC-2022.01
Record Dates: First submitted 2022-06-20; First posted 2022-06-27 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Radiofrequency ablation, High power, short duration: Radiofrequency ablation is an ablation modality that uses radiofrequency energy to create ablation lesions through heat. Patients that are scheduled for pulmonary vein isolation using radiofrequency ablation will be consented for study participation.
  Interventions: Device: Catheter ablation
- Ultra-low temperature cryo ablation: Ultra-low temperature cryo ablation is an ablation modality that uses nitrogen near its liquid-vapor critical point to create ablation lesions through ultra-low temperatures. Patients that are scheduled for pulmonary vein isolation using ultra-low temperature cryo ablation will be consented for study participation.
  Interventions: Device: Catheter ablation
- Pulsed field ablation: Pulsed field ablation is an ablation modality that uses short lived electrical fields to create ablation lesions through irreversible electroporation. Patients that are scheduled for pulmonary vein isolation using pulsed field ablation will be consented for study participation.
  Interventions: Device: Catheter ablation

INTERVENTIONS:
Device: Catheter ablation — An ablation catheter is introduced in the heart. Ablation is performed by applying ablation energy to the target tissue. The aim of ablation is to create an ablation lesion that does not conduct the electrical signals that induce or sustain the cardiac arrhythmia.

SUMMARY:
Ineffective ablation lesions can cause arrhythmia recurrence after catheter ablation for cardiac arrhythmia. Ablation lesions can be created with various ablation energy modalities. This study uses cardiovascular magnetic resonance imaging to evaluate the ablation lesion characteristics of radiofrequency ablation, ultra-low temperature cryo ablation, and pulsed field ablation. The ablation lesion characteristics of different energy characteristics will be compared. Additionally, arrhythmia recurrence and quality of life will be evaluated for the different energy modalities.

DETAILED DESCRIPTION:
Catheter ablation has become a cornerstone in the treatment of atrial fibrillation (AF). Typically, radiofrequency ablation (RFA) and cryoballoon ablation are used to perform pulmonary vein isolation (PVI). This treatment is effective in the majority of patients, but nevertheless 35% of patients have arrhythmia recurrence at 1-year follow up. These recurrence rates have been attributed to multiple factors, including ineffective ablation lesions, presence of non-pulmonary vein arrhythmia triggers, and disease progression.

Ineffective ablation lesions can cause arrhythmia recurrence through electrical reconnection. Electrical reconnection can occur when gaps are present in the ablation line due to non-durable, non-transmural or non-contiguous ablation lesions. Conventionally, ablation lesion assessment is performed using a redo electrophysiology study at three months post-ablation. During a redo electrophysiology study, a catheter is used to measure the local electrical signals to enable identification of sites with electrical reconnection. This method is effective but poses the patient to the procedural risks of these invasive measurements. Cardiovascular magnetic resonance (CMR) imaging may provide an alternative method for the evaluation of ablation lesions. Modern acquisition and post-processing techniques are under development and being used to image the atrial wall. These techniques may effectively visualize the fibrous tissue of ablation lesions, which enables a non-invasive method to characterize the lesions of catheter ablation.

To reduce arrhythmia recurrence caused by electrical reconnection, several novel ablation techniques have been developed in the last years. These novel ablation techniques can potentially reduce arrhythmia recurrence by enabling the creation of durable, transmural and contiguous ablation lesions. Novel ablation modalities include ultra-low temperature cryoablation (ULTC) and pulsed field ablation (PFA) that use near-critical nitrogen and pulsed electrical fields to create ablation lesions. The initial clinical outcomes of both ablation modalities are favorable, but little data are available on the ablation lesion characteristics. Additionally, novel techniques were developed to improve the procedural outcomes of RFA. High power, short duration (HPSD) RF energy applications cause more resistive and less conductive tissue heating compared to convention RFA, which results in more durable ablation lesions and less arrhythmia recurrence while safety outcomes are similar.

This study aims to use CMR to evaluate the ablation lesion characteristics of HPSD RFA, ULTC and PFA. This novel information can be used to quantitatively compare different ablation modalities. Furthermore, this study could contribute to our knowledge on ablation lesion formation, which may be used to further develop our ablation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years old)
* Paroxysmal or persistent atrial fibrillation, meeting criteria of the 2020 European Society of Cardiology Guidelines for diagnosis and management of atrial fibrillation
* Patients scheduled to undergo catheter ablation for cardiac arrhythmia using one of the following techniques: Radiofrequency ablation (High power, short duration), Ultra-low temperature cryo ablation, or Pulsed field ablation

Exclusion Criteria:

* Known (or suspected) allergic reaction to gadolinium
* Contraindications for MRI (such as claustrophobia, certain implants, devices, high body mass index).
* Pregnancy or breastfeeding
* Prior intervention in the left atrium (ablation or surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The studied population will be drawn from all patients that are scheduled for catheter ablation at the participating center.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Length of gaps in the ablation lesions | At 3 months follow up
  Cardiovascular magnetic resonance imaging is used to visualize the ablation lesion. If gaps are present in the ablation lesion, the length of the gaps is measured in millimeter.

SECONDARY OUTCOMES:
Number of gaps in the ablation lesion | At 3 months follow up
  Cardiovascular magnetic resonance imaging is used to visualize the ablation lesion. The number of gaps in the ablation lesion are counted.
Location of gaps in the ablation lesion | At 3 months follow up
  Cardiovascular magnetic resonance imaging is used to visualize the ablation lesion. If gaps are present in the ablation lesion, the location of the gaps is recorded.
Recurrence of atrial arrhythmia | Until 1 year of follow up
  Ambulatory rhythm monitoring will be performed at 3 and 12 months follow up to assess for recurrences of atrial arrhythmia (i.e. atrial fibrillation, atrial flutter, atrial tachycardia). Additionally, planned and symptom-driven electrocardiograms are assessed for atrial arrhythmia.
Atrial arrhythmia burden | Baseline, 3 and 12 months follow up
  Ambulatory rhythm monitoring will be performed at baseline, 3 and 12 months follow up to assess the atrial arrhythmia (i.e. atrial fibrillation, atrial flutter, atrial tachycardia) burden (proportion of time in atrial arrhythmia).
Atrial fibrillation related quality of life | Baseline, 3 and 12 months follow up
  A validated questionnaire (AFEQT) will be used to evaluate the atrial fibrillation related quality of life at baseline, 3 and 12 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas VA Boersma, MD, PhD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St. Antonius Hospital, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided